CLINICAL TRIAL: NCT05357469
Title: Innovative Treatment of Chemotherapy-Induced Painful Peripheral Neuropathy in Adolescents and Young Adults With Cancer: A Two Arm Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0657; NCI-2022-03832 (Other: NCI-CTRP-Clinical Trial Reporting Registry); 1R21CA256136-01A1 (NIH)
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Immediate St (Scrambler Therapy) (Experimental): Participant will start ST (Scrambler Therapy) treatment right away.
  Interventions: Device: Immediate St (Scrambler Therapy)
- Waitlist ST (Scrambler Therapy) (Experimental): Participant will start ST (Scrambler Therapy) treatment about 4 weeks after your Baseline Visit.
  Interventions: Device: Waitlist ST (Scrambler Therapy)

INTERVENTIONS:
Device: Immediate St (Scrambler Therapy) — Participant will receive Scrambler Therapy one (1) time a day, Monday through Friday, for up to 2 weeks (a total of 10 ST treatments).
  Arms: Immediate St (Scrambler Therapy)
Device: Waitlist ST (Scrambler Therapy) — Participant will receive Scrambler Therapy one (1) time a day, Monday through Friday, for up to 2 weeks (a total of 10 ST treatments).
  Arms: Waitlist ST (Scrambler Therapy)

SUMMARY:
To evaluate the efficacy and safety of Scrambler therapy (ST) for chemotherapy-induced painful peripheral neuropathy (CIPN), and the impact of ST on physical functioning and quality of life (QoL) in adolescents and young adults (AYA) cancer patients.

In this proposed study, we will conduct a two-arm prospective, randomized wait-list controlled clinical trial to investigate the effectiveness of ST on pain and CIPN in AYAs with cancer.

DETAILED DESCRIPTION:
Baseline Visit:

If you agree to take part in this study, you will have a Baseline Visit (a visit done before you begin receiving ST). At this visit:

You will have a physical exam. You will complete questionnaires about your symptoms, pain levels and how you think pain is affecting your life (such as your mood, ability to work, enjoyment of life, relationships with other people, and so on), quality of life, and your ability to walk and sleep. These questionnaires should take less than 30 minutes to complete. You will be asked about your pain medication use (including the name of the medications and how often you use them). You will complete a 6-Minute Walk Test. For this test, you will be asked to walk back and forth over a short distance as many times as you can for 6 minutes. This helps researchers measure your physical ability to walk and how well you can walk. You will have a sensory test to help researchers measure your touch sensation and your pain threshold for warm and cold temperatures. This test should take about 1 hour.

Study Groups and Scrambler Therapy:

After your Baseline Visit, you will be randomly assigned to 1 of 2 groups: Immediate ST or Waitlist ST. This is done because no one knows if one group is better, the same, or worse than the other. In Immediate ST, you will start ST treatment right away. In Waitlist ST, you will start ST treatment about 4 weeks after your Baseline Visit. You will have an equal chance (50/50) of being assigned to either group. The study staff will tell you which group you are in and when you will start treatment. You will receive Scrambler Therapy one (1) time a day, Monday through Friday, for up to 2 weeks (a total of 10 ST treatments). During each ST treatment session, about 2-10 pads, called electrodes, will be placed on your legs/feet or wrist/hands where you are experiencing pain, tingling, and/or numbness. A small electrical current will then be sent to the electrodes. At each session, you will receive the current for about 30-45 minutes.

Study Visits

Before each ST:

You will complete questionnaires about your pain levels and how you think pain is affecting your life, as well as the questionnaire about your ability to walk and sleep. These should take about 5-10 minutes to complete. copies You will be asked about your pain medication use.

At each ST session:

You will have a physical exam. You will have a sensory test.

Every week for 4 weeks after ST is complete, you will complete questionnaires about your pain levels and how you think pain is affecting your life, as well as the questionnaire about your ability to walk and sleep. You will also be asked about your pain medication use.

At Months 1, 2, and 3 after ST:

You will have a physical exam. You will have a sensory test. You will complete questionnaires about your pain levels and how you think pain is affecting your life, as well as the questionnaire about your ability to walk and sleep. You will be asked about your pain medication use.

At the Month 3 visit only:

You will complete the questionnaire about your quality of life. You will complete a 6 Minute Walk Test. Your participation in this study will be over after the 3-month visit

ELIGIBILITY:
Inclusion Criteria:

1. - Both genders aged 15-39 years
2. - Patients who have CIPN associated with at least moderate symptoms of pain (≥4 on a 0-10 scale) or neuropathy.
3. - Patients have had cancer and are not being actively treated,
4. - Patients who speaks English and able to complete questionnaires by themselves or with help from parents and/or nurses. Written informed consent will be obtained from adults (aged 18-39 years) or from parents/guardians of adolescents (aged 15-17 years) and assent will be obtained from adolescents (aged 15-17 years) under an Institutional Review Board (IRB)-approved protocol.

Exclusion Criteria:

1. - Inability to walk or stand without assistance (need for ambulatory-assist devices)
2. - Bone and/or central nervous system metastases that affect gait, walking and balance
3. - History of other known or unknown causes of acute or chronic neuropathic and/or no neuropathic pain conditions.
4. - Implanted intrathecal drug-delivery system or a spinal cord and/or peripheral nerve stimulator;

   a) a metal implant such as a cardiac pacemaker, automatic defibrillator, aneurysm clips, vena cava clips, or skull plate.
5. - History of epilepsy.
6. - Skin damage at the site of electrode placement; and i) prior ST treatment; j) Patients on pain medications for other than CIPN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The European Organization for Research and Treatment of Cancer ( EORTC-QLQ C30) | through study completion, an average of 1 year
  Five functional scales (physical, role, cognitive, emotional, and social); nine symptom scales (fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation, diarrhea, and financial difficulties); and a global health status/QoL. Based on 30 questions in total, the scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Salahadin Abdi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org